CLINICAL TRIAL: NCT02823119
Title: Mini-hysteroscopy Versus Conventional Office Hysteroscopy in Nulliparous Patients Undergoing Diagnostic Office Hysteroscopy: A Randomized Controlled Trial
Brief Title: Mini-hysteroscopy Versus Conventional Office Hysteroscopy in Nulliparous Patients Undergoing Office Hysteroscopy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Usama M Fouda, M.D, PhD, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hysteroscope size & pain
Record Dates: First submitted 2016-06-07; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Pain
Keywords: Mini-hysteroscopy; Office hysteroscopy; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mini-hysteroscopy (Experimental): A rigid 2.7-mm hysteroscope with a 30° forward oblique lens and an outer sheath diameter of 3.3 mm.
  Interventions: Device: Mini-hysteroscopy
- Conventional Office Hysteroscopy (Active Comparator): A rigid 2.9-mm hysteroscope with a 30° forward oblique lens and an outer sheath diameter of 5 mm
  Interventions: Device: Conventional Office Hysteroscopy

INTERVENTIONS:
Device: Mini-hysteroscopy — Hysteroscopy will be performed with the use of the non-touch technique (vaginoscopic approach). The investigators will use a rigid 2.7-mm hysteroscope with a 30° forward oblique lens and an outer sheath diameter of 3.3 mm. All of the procedures will be diagnostic.
  Arms: Mini-hysteroscopy
Device: Conventional Office Hysteroscopy — . Hysteroscopy will be performed with the use of the non-touch technique (vaginoscopic approach). The investigators will use a rigid 2.9-mm hysteroscope with a 30° forward oblique lens and an outer sheath diameter of 5 mm. All of the procedures will be diagnostic.
  Arms: Conventional Office Hysteroscopy

SUMMARY:
The aim of this study is to evaluate the effect of hysteroscope diameter on the pain experienced by nulliparous patients undergoing diagnostic office hysteroscopy.

DETAILED DESCRIPTION:
The results of the studies comparing the pain experienced by the patients undergoing conventional office hysteroscopy or mini-hysteroscopy were mixed. Several studies revealed that mini-hysteroscopy significantly reduced the procedure related pain and other studies revealed that the use of mini-hysteroscope was not associated with significant reduction in the procedure related pain. The aim of this study is to evaluate the effect of hysteroscope diameter on the pain experienced by nulliparous patients undergoing diagnostic office hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous patients

Exclusion Criteria:

* Parous patients, menopausal status, cervical pathology, and previous cervical surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | up to 30 minutes
  Intensity of pain assessed by the Visual Analog Scale (VAS)"

SECONDARY OUTCOMES:
Duration of procedure | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D, PhD, Study Director — Cairo University
Locations (1):
- Obstetrics and Gynecology Department,Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rullo S, Sorrenti G, Marziali M, Ermini B, Sesti F, Piccione E. Office hysteroscopy: comparison of 2.7- and 4-mm hysteroscopes for acceptability, feasibility and diagnostic accuracy. J Reprod Med. 2005 Jan;50(1):45-8. PMID 15730173